CLINICAL TRIAL: NCT05922904
Title: PET Adapted Brentuximab Vedotin and Pembrolizumab in Combination With Doxorubicin and Dacarbazine in Classic Hodgkin Lymphoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0492; NCI-2023-05028 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2023-06-20; First posted 2023-06-28 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease | interventions — Brentuximab Vedotin; Doxorubicin; pembrolizumab; Dacarbazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A: Pembrolizumab and Brentuximab +AD (Experimental)
  Interventions: Drug: Brentuximab vedotin; Drug: Doxorubicin Hydrochloride; Drug: Pembrolizumab; Drug: Dacarbazine
- Part B: De-Escalation (Experimental)
  Interventions: Drug: Brentuximab vedotin; Drug: Doxorubicin Hydrochloride; Drug: Pembrolizumab; Drug: Dacarbazine
- Part C: Standard Risk Arm (Experimental)
  Interventions: Drug: Brentuximab vedotin; Drug: Doxorubicin Hydrochloride; Drug: Pembrolizumab; Drug: Dacarbazine

INTERVENTIONS:
Drug: Brentuximab vedotin — Given by IV (vein)
Drug: Doxorubicin Hydrochloride — Given by IV (vein)
  Other Names: Adriamycin PFS®; Adriamycin RDF™; Adriamycin®; Rubex®
Drug: Pembrolizumab — Given by IV (vein)
  Other Names: SGN-35; Adcetris
Drug: Dacarbazine — Given by IV (vein)
  Other Names: DTIC-Dome®

SUMMARY:
To learn about the effects of brentuximab vedotin and pembrolizumab in combination with doxorubicin and dacarbazine when given to patients who have Stage II cHL with bulky mediastinal disease or advanced cHL (Stage III or IV) and who have not received treatment for the disease.

DETAILED DESCRIPTION:
Primary Objectives:

● To assess the complete response (CR) rate at the end of therapy (EOT) with Brentuximab vedotin and pembrolizumab, doxorubicin and dacarbazine in subject with previously untreated stage II bulky mediastinal disease or advanced stage cHL.

Secondary Objectives:

* To assess the safety of BvP+AD
* To assess the complete remission rate at interim PET (CR iPET)
* To assess the overall response rate (ORR)
* To assess the duration of response (DOR)
* To assess the duration of complete response (DOCR)
* To assess event-free survival (EFS)
* To assess progression free survival (PFS)
* To assess overall survival (OS)

ELIGIBILITY:
Inclusion Criteria:

1. Treatment-naïve, HL subjects with Ann Arbor stage III, IV, or stage II with bulky disease (>10 cm).
2. Histologically confirmed cHL according to the current World Health Organization Classification (nodular sclerosis, mixed cellularity, lymphocyte rich, lymphocyte depleted, classical HL, or not otherwise specified). a. Subjects enrolling must submit a tumor block for analysis. Availability of tissue must be confirmed prior to enrollment.
3. Bidimensional measurable disease as documented by PET/CT or CT imaging. Must have at least one lesion >15 mm (1.5 cm) in the longest diameter on cross-sectional imaging, measurable in 2 perpendicular dimensions on CT (or MRI), and FDG avid by PET.
4. Age 18 years or older.
5. An Eastern Cooperative Oncology Group (ECOG) performance status zero, or one.
6. Subjects of childbearing potential must have a negative serum or urine beta human chorionic gonadotropin (β-hCG) pregnancy test result within 7 days prior to the first dose of brentuximab vedotin. Subjects with false positive results and documented verification that the subject is not pregnant are eligible for participation. Subjects of non-childbearing potential are those who are postmenopausal >1 year or who have had a bilateral oophorectomy or hysterectomy.
7. If sexually active in a way that could result in pregnancy, subjects of childbearing potential must agree to use 2 effective contraception methods during the study and for 7 months following the last dose of study drug. Subjects who can father children and have partners of childbearing potential must agree to use 2 effective contraception methods during the study and for 7 months following the last dose of study drug. Subjects who can father children must also be willing to refrain from sperm donation during this time.
8. The subject or the subject's legally acceptable representative must provide written informed consent. Cognitive ability will be assessed according to policy CLN0547.
9. The following baseline laboratory data:

   * absolute neutrophil count ≥1500/μL unless there is known HL marrow involvement
   * platelet count ≥75,000/μL
   * serum bilirubin ≤1.5 x upper limit of normal (ULN) or ≤3 x ULN for subjects with Gilbert's disease
   * estimated glomerular filtration rate (GFR) ≥30 mL/min/1.73 m2 using the Modification of Diet in Renal Disease (MDRD) study equation as applicable
   * alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3 x ULN or ≤5 x ULN if there is documented hepatic involvement of HL
   * hemoglobin ≥8 g/dL

Exclusion Criteria:

1. Nodular lymphocyte predominant HL.
2. History of another malignancy within 3 years before the first dose of study drug or any evidence of residual disease from a previously diagnosed malignancy. Exceptions are malignancies with a negligible risk of metastasis or death (e.g., 5-year OS ≥90%), such as adequately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, localized prostate cancer, ductal carcinoma in situ, or Stage I uterine cancer. Subjects with nonmelanoma skin cancer, localized prostate cancer, or carcinoma in situ of any type are not excluded if they have undergone complete resection.
3. Prior immunosuppressive chemotherapy, therapeutic radiation, or any immunotherapy (e.g., immunoglobulin replacement, other monoclonal antibody therapies) within 4 weeks of first study drug dose, unless underlying disease has progressed on treatment.
4. Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, or anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways.
5. Active cerebral/meningeal disease related to the underlying malignancy, including signs or symptoms of progressive multifocal leukoencephalopathy (PML) or history of PML. Subjects with a history of cerebral/meningeal disease related to the underlying malignancy are allowed if prior CNS disease has been treated.
6. Any active Grade 3 or higher (per the National Cancer Institute's Common Terminology Criteria for Adverse Events [NCI CTCAE] Version 4.03) viral, bacterial, or fungal infection within 1 week prior to the first dose of study drug. Routine antimicrobial prophylaxis is permitted.
7. Current therapy with other systemic anti-neoplastic or investigational agents.
8. Planned consolidative radiotherapy.
9. Active interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected drug-related pulmonary toxicity.
10. Grade 3 or higher pulmonary disease unrelated to underlying malignancy.
11. Idiopathic interstitial pneumonia or diffusing capacity of the lung for carbon monoxide (adjusted for hemoglobin) <50% predicted.
12. Documented history of a cerebral vascular event (stroke or transient ischemic attack), unstable angina, myocardial infarction, or cardiac symptoms consistent with New York Heart Association Class III-IV within 6 months prior to their first dose of brentuximab vedotin. See Appendix E
13. Subjects with Child-Pugh class B or C hepatic impairment.
14. Other serious underlying medical condition that, in the opinion of the investigator, would impair the subject's ability to receive or tolerate the planned treatment and follow-up.
15. Symptomatic neurologic disease compromising normal activities of daily living or requiring medications. See Appendix G
16. Grade 2 or higher peripheral sensory or motor neuropathy at baseline.
17. Left ventricular ejection fraction <45% or symptomatic cardiac disease (including symptomatic ventricular dysfunction, symptomatic coronary artery disease, and symptomatic arrhythmias), or previous treatment with complete cumulative doses of doxorubicin or other anthracyclines.
18. Subjects with acute or chronic graft-versus-host-disease (GvHD) or receiving immunosuppressive therapy as treatment for or prophylaxis agent against GvHD.
19. Previous treatment with brentuximab vedotin.
20. Known history of hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection.
21. Known to be positive for human immunodeficiency virus (HIV).
22. Subjects who are pregnant or breastfeeding.
23. Known hypersensitivity to any excipient contained in the drug formulation of brentuximab vedotin, any component of AD, pembrolizumab, doxorubicin, dacarbazine, filgrastim, or pegfilgrastim.
24. Treatment with botanical preparations (e.g., herbal supplements, traditional Chinese medicines) intended to treat the disease under study within 2 weeks prior to treatment.
25. Subjects who have received a live or attenuated vaccine within 30 days prior to treatment.
26. Subjects with an active autoimmune disease or any other condition requiring systemic treatment with either corticosteroids within 7 days (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 30 days of starting treatment. Inhaled or topical steroids, and adrenal replacement steroid doses >10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease. a. Subjects with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
27. Subjects who received organ transplant or allogeneic stem cell transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-12-14 (Actual); Primary Completion 2027-10-30 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0 | through study completion; an average of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Hun Lee, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Kreuzberger N, Goldkuhle M, von Tresckow B, Kobe C, Sickinger MT, Monsef I, Skoetz N. Positron emission tomography-adapted therapy for first-line treatment in adults with Hodgkin lymphoma. Cochrane Database Syst Rev. 2025 Mar 26;3(3):CD010533. doi: 10.1002/14651858.CD010533.pub3. PMID 40135712
- See also: M D Anderson Cancer Center — http://www.mdanderson.org